CLINICAL TRIAL: NCT05403684
Title: Impact of Hindmilk on Weight Gain Among Moderate to Very Preterm Infants in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Chiesi Foundation (Unknown)
Responsible Party: Principal Investigator, Albert Manasyan, MD, MPH, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300007476
Record Dates: First submitted 2022-05-23; First posted 2022-06-03 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Postnatal Growth Restriction
Keywords: breastmilk; hindmilk; high-volume breastfeeding; postnatal growth restriction; preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The proposed study is a non-blinded randomized controlled trial with a 1:1 parallel allocation of infants to higher-volume feedings (200-240 ml/kg/day) or usual-volume feedings (140-180 ml/kg/day) using computer-generated random-block sequences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual-volume breastfeeding (UV Group) (No Intervention): Infants will receive cup-feeding (to standardize the volume at each feeding) per standard of care guidelines (SOC: 140-180 mL/kg/day) with volumes adjusted for weight and infant age.
- High-volume breastfeeding (HV Group) (Experimental): Along with SOC volume provided via cup-feeding, the mother will continue to express and feed the baby hind-milk reaching 240 mL/kg/day with volumes adjusted for weight and infant age (200-240 ml/kg/day).
  Interventions: Other: High-volume breastmilk

INTERVENTIONS:
Other: High-volume breastmilk — Preterm infants will be given high-volume breastmilk
  Arms: High-volume breastfeeding (HV Group)

SUMMARY:
The primary hypothesis is that very preterm infants between 28 0/7 to 31 6/7 weeks with a birth weight from 1000-1999 grams allocated to the HV breastmilk group (200-240 mL/kg/day) until hospital discharge or 40 weeks' post-menstrual age (PMA), whichever comes first, will have increased growth velocity compared to those given UV breastmilk (140-180 mL/kg/day).

DETAILED DESCRIPTION:
The proposed study is a non-blinded randomized controlled trial with a 1:1 parallel allocation of infants to higher-volume feedings (200-240 ml/kg/day) or usual-volume feedings (140-180 ml/kg/day) using computer-generated random-block sequences. The study will enrol a total of 214 study participants including 190 preterm infants randomized controlled trial of HV feedings and 24 mothers of enrolled infants and healthcare workers for in-depth interviews. We will also screen mothers to study participants for postpartum depression using the Edinburgh Postnatal Depression Scale (EPDS) screening tool.

Study aims are:

Aim 1: To evaluate the impact of high volume (HV) feedings using additionally expressed milk at the end of feeding (hind-milk) vs usual volume (UV) feedings on growth velocity from birth to discharge or 40 weeks' PMA, whichever comes first, among very preterm infants.

Through a 1:1 randomization, the study will enrol 190 preterm infants weighing between 1,000g - 1,999g in both study arms and follow them until hospital discharge or 40 weeks' PMA, whichever comes first.

Aim 2: To evaluate the impact of HV vs UV breastfeeding until 40 weeks' PMA on all-cause neonatal mortality and morbidity (including sepsis, NEC, intestinal perforation, and hypoglycaemia).

All study participants (n=190) will be until 40 weeks' PMA to estimate its impact on all-cause neonatal mortality and morbidity.

Aim 3: To characterize the acceptability, feasibility, and feeding tolerance among HV breastfeeding women and their infants at the hospital and its feasibility by healthcare workers.

A total of 24 mothers and healthcare workers will be interviewed through in-depth interviews (IDIs) to better understand the acceptability of this intervention by the feeding mothers, the feeding tolerance by their newborns, and the feasibility of the same by the healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Between 28 0/7 to 31 6/7 weeks of age or weighing between 1000-1999 grams,
* Admitted to the UTH NICU within 24 hours after birth, and
* Infants who have reached feeding volume ≥120 mL/kg/day at time of randomization

Exclusion Criteria:

* Who are deemed unstable by the neonatologist,
* With necrotizing enterocolitis or intestinal perforation
* Known gastrointestinal malformations,
* Major malformations or congenital anomalies, and
* Whose parents do not provide informed consent

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Weight gain | Baseline up to 40 weeks PMA.
  Average change in weight between enrolment (baseline) up to 40 weeks post-menstrual age (PMA) or hospital discharge, whichever comes first.

SECONDARY OUTCOMES:
Head circumference | Baseline up to 40 weeks PMA.
  Average change in head circumference (in centimetres using measuring tape) between enrolment (baseline) and 40 weeks post-menstrual age (PMA) or hospital discharge, whichever comes first.
Mid-arm circumference | Baseline up to 40 weeks PMA.
  Average change in mid-arm circumference (in centimetres using measuring tape) between enrolment (baseline) and 40 weeks post-menstrual age (PMA) or hospital discharge, whichever comes first.
Length | Baseline up to 40 weeks PMA.
  Average change in length (in centimetres using measuring tape) between enrolment (baseline) and 40 weeks post-menstrual age (PMA) or hospital discharge, whichever comes first.
Length of hospital stay | Baseline up to 40 weeks PMA.
  Average change in length of hospital stay between enrolment (baseline) and 40 weeks post-menstrual age (PMA) or hospital discharge, whichever comes first.
Characterise acceptability, feasibility, and feeding tolerance by breastfeeding women and their infants | Through study completion, on average 8 weeks after enrolment
  To characterize the acceptability, feasibility, and feeding tolerance among HV breastfeeding women and their infants at the hospital.
Characterise feasibility of HV breastfeeding by healthcare workers (HCWs) | Through study completion, on average 8 weeks after enrolment
  To characterize the feasibility of HV breastmilk by mothers to the infants (patients) by HCWs

OTHER OUTCOMES:
Neonatal mortality | 28 days after birth
  Newborn status at 28 days after birth
Weight at 40 weeks PMA | 40 weeks PMA
  For infants discharged prior to 40 weeks PMA, their birthweight will be taken at 40 weeks PMA during study exit.
Postpartum Depression | 6-8 weeks postnatal
  Maternal postpartum depression at at 6-8 weeks postnatally using Edinburgh Postnatal Depression Scale screening tool (scale ranges from 0-30, with 11+ indicative of depressive symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Carlo, MD, Study Chair — University of Alabama at Birmingham; Colm Travers, MD, Study Director — University of Alabama at Birmingham; Albert Manasyan, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared upon a reasonable request to the study PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for sharing following publication of study findings (or during submission for publication if requested by the journal)
Access Criteria: Following a reasonable request to the study PI.